CLINICAL TRIAL: NCT06695871
Title: Effect of Patient Navigation-based Health Management Model on Quality of Life and Sexual Function After LEEP in Patients With Cervical Lesions
Brief Title: Research on the Application of Patient Navigation-based Management Model of Patients After LEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Ren Wenhui, Assistant research fellow, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024PHB398-001; MBZX0102024007 (Other Grant/Funding Number: Beijing Research Association for Chronic Diseases Control and Health Education)
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cervical Intraepithelial Neoplasias
Keywords: Loop electrosurgical excision procedure; Patient navigation; Quality of life; Sexual function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The routine clinical outpatient follow-up protocol was implemented, and a postoperative rehabilitation health manual was provided to patients the day following LEEP surgery. Outpatient evaluations were subsequently conducted at 1 month, 3 months, and 6 months post-surgery.
- Intervention group (Experimental): A postoperative rehabilitation health manual was provided to patients the day following LEEP surgery. The nursing team, possessing over one year of clinical experience in gynecological nursing and psychological counseling, collaborated with clinicians to deliver health consultation services. They conducted in-person consultations lasting 10-15 minutes during routine outpatient follow-ups at 1, 3, and 6 months post-surgery. Patients were assessed based on the challenges encountered in postoperative rehabilitation and sexual life, and tailored guidance services were administered. Additionally, online counseling and guidance services were offered at 2, 4, or 5 months following surgery.
  Interventions: Other: Patient navigation-based health management

INTERVENTIONS:
Other: Patient navigation-based health management — A patient navigation-based health management model for individuals with cervical lesions post-LEEP procedure, encompassing healthcare consultation services, personalized health guidance, and routine follow-up assessments.
  Arms: Intervention group

SUMMARY:
Cervical cancer poses a significant threat to women's health and is a crucial public health issue. Early detection and treatment of cervical lesions and standardized management have emerged as essential pillars in the Global Cervical Cancer Elimination. The loop electrosurgical excision procedure (LEEP) is widely employed as a preferred approach for the diagnosis and treatment of precancerous cervical lesions and early invasive cervical cancer. Patients with high-grade cervical lesions are more prone to experiencing sexual dysfunction and psychological disorders after LEEP, attributed to the unique surgical site, physiological alterations, and psychological stress during the postoperative recovery process, thereby adversely affecting their quality of life. Currently, there is a shortage of research evidence regarding targeted intervention measures and long-term effect evaluations for sexual function quality and quality of life after LEEP for cervical lesions. In recent years, the health management model based on patient navigation has evolved into a novel modality for facilitating comprehensive tumor prevention and control. However, its effect in managing cervical lesions has yet to be comprehensively assessed. Therefore, we will design a randomized controlled trial to evaluate the impact of a patient navigation-based health management model on quality of life and sexual function after LEEP in patients with cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 25 and 50 years;
* LEEP will be conducted following clinical evaluation;
* No intention to conceive within the subsequent year;
* Proficiency in utilizing social media platforms, such as WeChat, is required;
* Patients must be capable of providing informed consent to participate in the study and willing to engage in long-term follow-up.

Exclusion Criteria:

* Individuals who are widowed, separated, or experiencing atypical sexual activity due to reasons related to their spouse.
* Presence of genital tract malformations.
* A history of neurological disorders, such as stroke or epilepsy, or a history of psychiatric conditions, such as depression.
* Patients with other significant illnesses that could impact the long-term follow-up of the study.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | six months after LEEP
  The quality of life six months post-surgery was assessed using 36-Item Short Form Survey.

SECONDARY OUTCOMES:
Sexual function index | before LEEP, three months after LEEP, and six months after LEEP
  The Chinese version of the Female Sexual Function Index was used to evaluate the sexual function index at three time points: before LEEP, three months after LEEP, and six months after LEEP.
Anxiety | before LEEP, three months after LEEP, and six months after LEEP
  Anxiety symptoms were assessed using the Self-Rating Anxiety Scale at three-time points: before LEEP, three months after LEEP, and six months after LEEP.
Quality of Life | before LEEP and three months after LEEP
  The quality of life was assessed using 36-Item Short Form Survey.
Depression | before LEEP, three months after LEEP, and six months after LEEP
  Depression symptoms were assessed using the Self-Rating Anxiety Scale at three time points: before LEEP, three months after LEEP, and six months after LEEP.
Vaginal discharge | three and six months after LEEP
  Patient-reported alterations in the volume, color, and odor of vaginal secretions.
Recurrence rates | three and six months after LEEP
  The recurrence of cervical lesions at three and six months post-surgery was evaluated using high-risk HPV testing, cytology test, and histopathological examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China